CLINICAL TRIAL: NCT00670163
Title: Comunidades Positivas and Enhanced Partner Therapy in Peru
Brief Title: Effectiveness of Community-Level Behavioral and Biomedical Interventions for Reducing HIV/STIs in Men in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas J. Coates, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01MH078752 (NIH); R01MH078752 (NIH); DAHBR 9A-ASGP
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections; Sexually Transmitted Infections
Keywords: Men Who Have Sex With Men
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Homosexuality | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participating community will provide Comunidades Positivas plus enhanced partner therapy.
  Interventions: Behavioral: Enhanced Partner Therapy (EPT); Behavioral: Communidades Positivas (CPOS)
- 2 (Experimental): Participating community will provide enhanced partner therapy alone.
  Interventions: Behavioral: Enhanced Partner Therapy (EPT)
- 3 (Experimental): Participating community will provide Comunidades Positivas alone.
  Interventions: Behavioral: Communidades Positivas (CPOS)
- 4 (Active Comparator): Participating community will provide standard of care.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Enhanced Partner Therapy (EPT) — EPT, a biomedical intervention, is designed to reduce the rate of sexually transmitted infection (STI) reinfection and, therefore, incident STIs. Men who have sex with men (MSM) with incident STIs will be given partner treatment packets that contain informational brochures, reference cards, prophylactic medications, and condoms for their sexual partners.
  Other Names: EPT
  Arms: 1; 2
Behavioral: Communidades Positivas (CPOS) — The behavioral intervention, CPOS, is based on a combination of social-action theory and diffusion of innovation and is designed to reduce the frequency of unprotected sex with nonprimary partners. In CPOS, MSM who are recognized by their peers as leaders will be trained to implement a community center that provides information, support, and empowerment to MSM, their friends, and partners. CPOS will include a training program of at least 14 sessions. During these sessions, MSM leaders will be provided with information about HIV/STIs and their prevention and ways to strengthen leadership skills. The 2-hour group sessions will occur two times a week for 7 weeks. While the training sessions are underway, MSM leaders will be asked to work with community leaders to form a community center from which they will carry out HIV/STI prevention and promotion of sexual health activities for 18 months.
  Other Names: CPOS
  Arms: 1; 3
Behavioral: Standard Care — Standard care will consist of usual care for STIs.
  Arms: 4

SUMMARY:
This study will evaluate the effectiveness of community-level behavioral and biomedical interventions, each alone and combined, in reducing sexual risk behavior and HIV/sexually transmitted infections in Peruvian men who have sex with men.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs), including HIV, are among the most significant public health concerns worldwide. Although common across all groups of people, STIs have had a considerable impact among men who have sex with men (MSM). Particularly, in Peru, which accounts for about 6% of the estimated HIV infections in Latin America, HIV and STIs are highly concentrated in the MSM population.

Both behavioral and biomedical interventions are needed to provide education about the health risks associated with unprotected sex and to help those with STIs seek treatment. Communidades Positivas (CPOS) (Spanish for "Positive Communities") is a behavioral intervention designed to reduce the frequency of sexual activity with nonprimary partners. Enhanced partner therapy (EPT) is a biomedical intervention designed to provide treatment to partners who may become or already are infected with an STI and to thereby reduce the rate of reinfections. When implemented individually or together at a community level, these interventions may be effective in preventing HIV/STI transmission in MSM. This study will evaluate the effectiveness of community-level CPOS and EPT, each alone and combined, in reducing sexual risk behavior and HIV/STIs in Peruvian MSM.

Participation in this study will last 18 months. A total of 24 communities will be assigned randomly to 1 of 4 different treatment groups:

* Communities in Group 1 will provide CPOS plus EPT to MSM.
* Communities in Group 2 will provide CPOS alone to MSM.
* Communities in Group 3 will provide EPT alone to MSM.
* Communities in Group 4 will provide standard care to MSM.

Within each community, a select number of MSM will be evaluated at various points during the study. The initial evaluation visit will occur prior to any treatment and will include an interview, counseling, and HIV/STI testing. The interview will involve questions about health and community, including topics such as sexual activities, views on health problems, use of alcohol and drugs, use of health care services, and attitudes about people with HIV or AIDS. Counselors will then provide information about contracting and preventing HIV/STIs and will ask questions about STI symptoms. Finally, HIV/STI testing will be conducted and throat and anal swabs will be collected. Two weeks after the initial evaluation, MSM will receive their test results, and if positive for HIV or any STIs, they will receive appropriate referrals, services, and treatments. They will also receive the specific treatment to which their community was assigned and will be asked additional questions concerning the treatment of their partners, if applicable. The remaining evaluations, which will repeat assessments from the initial evaluation, will occur at months 9 and 18.

Standard care will include the care that has been established by the Peruvian national guidelines for managing HIV and STIs. In EPT, MSM will be encouraged to pass along to their recent partners packets that contain informational brochures, reference cards, prophylactic medications, and condoms. In CPOS, MSM who are recognized by their peers as leaders will be trained to implement a community center that provides information, support, and empowerment to MSM, their friends, and their partners.

ELIGIBILITY:
Inclusion Criteria:

For MSM evaluation group:

* Anatomically male at birth (by self-report)
* Lives in study barrio OR works in study barrio OR socializes in study barrio (present at least 3 times per week)
* Anal or oral sexual intercourse with another male in the 12 months before study entry
* Stated preference for sexual relations with males

For CPOS group:

* Self-identifies as a man who has sex with men

Exclusion Criteria:

For all participants:

* Imminent plans to move away from the study barrio for the duration of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 718 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of STIs | Measured at Month 18

SECONDARY OUTCOMES:
Rates of unprotected intercourse with nonprimary partners | Measured at Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Coates, PhD, Principal Investigator — The University of California, Los Angeles (UCLA)
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Lima Province, Peru

REFERENCES:
- [Derived] Leon SR, Segura ER, Konda KA, Flores JA, Silva-Santisteban A, Galea JT, Coates TJ, Klausner JD, Caceres CF. High prevalence of Chlamydia trachomatis and Neisseria gonorrhoeae infections in anal and pharyngeal sites among a community-based sample of men who have sex with men and transgender women in Lima, Peru. BMJ Open. 2016 Jan 6;6(1):e008245. doi: 10.1136/bmjopen-2015-008245. PMID 26739719